CLINICAL TRIAL: NCT06514547
Title: Vaccine Immunity and Inflammation in the Aging Person Living With HIV
Acronym: VIVID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anne Frosch, Principal Investigator, Hennepin Healthcare Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FY2024-738; 1R01AG084437-01A1 (NIH)
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections; Age
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: 1) Some participants will receive this vaccine as part of routine clinical care, and we will coordinate our study visits based on the receipt of that vaccine. 2) Some participants will receive this vaccine outside of the Centers for Disease Control and Prevention recommended schedule, but as in accordance with FDA approved use and 3) Some participant who are receiving this vaccination outside of current FDA approval for a single dose in those above 18 by receiving a second dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pneumococcal Vaccination (Experimental): All participants will receive a pneumococcal vaccine.
  Interventions: Biological: Conjugate Pneumococcal Vaccine 20 (PCV20)

INTERVENTIONS:
Biological: Conjugate Pneumococcal Vaccine 20 (PCV20) — Vaccine
  Other Names: Prevnar20

SUMMARY:
This study will track immune responsiveness to conjugate pneumococcal vaccines over time to help determine how long protection from this vaccine lasts in individuals with chronic medical conditions (in this study - HIV) and with age.

DETAILED DESCRIPTION:
Persons living with HIV (PLWH) are at increased risk of chronic inflammation and the associated adverse health outcomes. There is considerable evidence that chronic inflammatory conditions like metabolic disease and autoimmune disorders as associated with weakened vaccine responses and existing vaccine studies in PLWH do not adequately sample older individuals who are disproportionately affected by this "inflammaging." We hypothesize the effect of age on poor vaccine responses is greater among PLWH given the additional burdens of HIV driven inflammation. The overall project goal is to examine this premise by measuring the impact of HIV status, age, and chronic immune activation on conjugate pneumococcal vaccine responses. We will study acute (30 day) and longer-term (2 year) immune responses following PCV vaccination, among a cohort of participants including 4 groups: a) older PLWH, age ≥50 (n=100), b) older HIV uninfected controls, age ≥50 (n=50), c) younger PLWH, age <50 (n=50), d) younger HIV uninfected controls, age <50 (n=50). With these cohorts, we will 1) Comprehensively characterize the impact of HIV and age on the immunogenicity of conjugate pneumococcal vaccination by longitudinally tracking adaptive vaccine-specific antibody, B cell and cluster of differentiation 4 T cell responses. We will compare these responses by age and HIV status. We will also 2) Determine the influence of chronic inflammation on vaccine-specific immunity among PLWH across the adult lifespan by measuring the associate between vaccine immunity and biomarkers of chronic inflammation. This project will provide valuable knowledge on how HIV and age influence vaccine immune responses with the hope of informing vaccine development and schedule to optimize the long-term health of persons living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* HIV Diagnosis
* On Antiretroviral Therapy with HIV Viral Load<200 within last year

Exclusion Criteria:

* Other significant immunosuppressing condition
* Age< 18 years
* Pregnancy (at enrollment)
* Contraindication to pneumococcal vaccination
* Known contraindication to non-clinical blood draws (severe anemia last hemoglobin <8g/dl)
* Subjects who, in the opinion of the Investigator, may be non-adherent to study schedules or procedures.
* Adults unable to consent
* Individuals with impaired ability to consent
* Incarceration at time of enrollment

Controls inclusion criteria:

* Age>=18 years
* HIV Ag-Ab test negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 30 days and 2 years
  Evaluate the impact of HIV status on pneumococcal vaccine immunogenicity and durability as measured pneumococcal-specific Ab concentration, memory B cell responses (frequency and phenotype) and CD4 T cell responses (frequency and phenotype) at an acute (primary comparison) and memory (secondary comparison) post-vaccination timepoints.

SECONDARY OUTCOMES:
Secondary objective | 30 days and 2 years
  Explore the impact of advanced age on pneumococcal vaccine immunogenicity and durability in PLWH. This will be evaluated by evaluating the relationship of age and pneumococcal-specific Ab concentration, memory B cell responses (frequency and phenotype) and CD4 T cell responses (frequency and phenotype) at acute and memory timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided